CLINICAL TRIAL: NCT02924207
Title: Electronic Decision Support for Intervention in Poorly Controlled Type 2 Diabetes
Acronym: PATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Elizabeth Healthcare (Other)
Collaborators: PATH Decision Support Software, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6/2016-018
Record Dates: First submitted 2016-09-29; First posted 2016-10-05 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Path Electronic decision support arm
  Interventions: Other: PATH electronic decision support tool

INTERVENTIONS:
Other: PATH electronic decision support tool — PATH, a clinical decision support tool for Type 2 Diabetes, was developed based on patient impact of efficacy, cost, implementation difficulty, comorbidities, side effects, and evidence based pleiotropic benefit. Drug efficacy was estimated using published clinical data for agents, both in terms of placebo controlled trials and head-to-head studies. Additional information regarding interventions was added with regard to FDA package inserts as well as large post marketing studies. Cost impact of intervention was described in terms of patient's estimated copay drawn from insurance plan as well as average retail price.

SUMMARY:
To determine the impact of an electronic decision support tool on physician decision making and patient outcomes for the treatment of poorly controlled diabetes mellitus. Primary endpoint will measure change in hemoglobin A1c. Secondary endpoints will examine cost of therapy and patient satisfaction with therapy. Study hypothesis is that use of the PATH decision tool will produce greater reduction overall in measurements of hemoglobin A1c in patients who participate and follow the PATH decision tool than patients who elect not to follow the PATH decision tool. PATH decision tool will provide more cost effective solutions for management of diabetic medication than current methods.

DETAILED DESCRIPTION:
1. Patients of selected St. Elizabeth Physicians Primary Care Physicians without a new intervention related to the management of the patient's diabetes in the last 3 months may be contacted via telephone by research staff.
2. During the telephone call, patients will be offered the opportunity to manage their diabetic medication by following the PATH decision tool, explaining that PATH is a computer program which finds a balance between low cost and high effectiveness. If participation is elected, informed consent will be mailed with a follow up phone call from staff, or an informed consent will be signed at their upcoming primary care office visit. Some patients may be approached during their office visit, without a prior phone call. Patients who do not have an eligible hemoglobin A1c on file, but are expecting to have an eligible hemoglobin A1c value on an upcoming blood test may consent prior to the blood test. If the hemoglobin A1c comes back >=7.0, the patient will continue following protocol. If the hemoglobin A1c comes back <7.0, the patient will be categorized as a screen failure, but will remain eligible for later enrollment. If the patient becomes eligible and is later enrolled, the patient will be assigned a new study ID number.

   i) If a patient elects not to participate, the reason for not participating may be recorded in the screening log. As part of the standard of care, patients not selecting the study will be offered an appointment outside the study to address their poorly controlled diabetes.

ii) If a patient elects to participate and a hemoglobin A1c has not been drawn in the last 3 months, one will be ordered through their insurance as part of the standard of care, to be used as the baseline hemoglobin A1c for Path calculations.

3. Patients who agree to participate maybe contacted by telephone by a licensed provider (MD or ARNP) who will enter non identifiable data from the patient's chart into the PATH decision support software. Information will be gathered from the Epic EHR and the questionnaire found on Article #2. This questionnaire may be completed by the patient, or by staff during patient interview. Some patients may complete this process during their scheduled office visit.

i) Study specific items will be recorded as illustrated in Article #4 ii) Time spent populating the data will be recorded, as part of the secondary analysis.

4. Patient and provider will discuss options on the telephone or during the office visit, and will further customize regimen selections while discussing risks and benefits. Once a regimen is selected, the score and content of the regimen will be recorded by the provider.

i) Regimen selected will be classified by "partial recommendation, full recommendation, alternate recommendation, or "no action" in relation to the options presented by the PATH program. --> final score of the course of action will be calculated and recorded.

i. Definitions:

1. Full recommendation: the regimen selected is the exact regimen shown in PATH, with no additions or deletions.
2. Subset recommendation: the regimen selected is a subset of a regimen shown in PATH (i.e., with one or more deletions), with no additions.

   1. Example: PATH recommends the regimen (A, B, C, D)
   2. Valid subset regimens would include (A, B, C), (B, C, D), (A, B), and (A), among others.
3. Superset recommendation: the regimen selected contains all of the elements of one regiment recommended by PATH, plus at least one other therapy.

   1. Example: PATH recommends the regimen (A, B, C)
   2. A valid superset recommendation would be (A, B, C, Exercise).
4. Alternate recommendation: Any other combination of additions and deletions from a PATH recommended regimen.
5. No action: No regimen was selected.

5. Manufacturer Discount coupons will be offered and mailed if applicable as part of the normal procedures of the primary care office.

i) Mailed coupons will be documented in the participant's study chart.

6. If Path is completed over the phone, the patient will be offered immediate "in person" follow up (traditional visit) to review the changes. As this is appropriate to the treatment of diabetes, traditional CPT billing will be used and the in-person visit will be billed to insurance as part of standard of care.

i) Patient's choice to participate in a traditional office visit will be recorded in the participant's study chart.

7. Follow up visit or phone call will be scheduled at 3 months (+/- 30 days) with repeat hemoglobin A1c, following the standard of care for the treatment of diabetes. The 3 months (+/- 30 days) follow up window will be calculated from the date patients are informed of their new medication regimen. During this visit, diabetes evaluation will follow the standard of care including adherence, efficacy, and adverse events. Adverse events will be categorized through the "drug intolerance" and "comorbidities" section of the PATH software. See Article #6 i) Type of follow up will be recorded ("phone follow up, live follow up, no follow up"). Reason for no follow up will also be documented.

ELIGIBILITY:
Inclusion Criteria:

* Patient under the care of a primary care physician within St. Elizabeth Physicians
* >=18 years of age
* Diagnosis of Type 2 Diabetes for at least 6 months
* Hemoglobin A1c values of >= 7.0 (drawn within the last year).

Exclusion Criteria:

* Type 1 Diabetes, Secondary Diabetes, Gestational Diabetes or LADA (presence of anti-GAD, IA-2, C-Peptide <0.5)
* Participant is currently or intended to start hemodialysis or peritoneal dialysis during the course of the study.
* Chronic or planned systemic glucocorticoid use
* Scheduled prandial insulin therapy (premix and basal okay)
* Other health threatening disease state at investigator's discretion
* Potential participant is unable to fully comprehend the risks of study participation or comply with study procedures.
* New diabetes intervention in the last 3 months (change in diabetes medication or dosage)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-09; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
change in hemoglobin A1c from baseline | 1 year
  change in hemoglobin A1c from baseline

SECONDARY OUTCOMES:
change in patient's perception of cost of diabetes medicine and side effects | 1 year
  At baseline and 3 month follow up visits, patients will be asked to rate affordability of their medications on a scale of 1 to 10. Subjects will also be asked to rate their satisfaction on a scale of 1 to 10.
actual cost and change in frequency of drug side effects | 1 year
  The actual change in the cost of the subjects medication will be recorded and compared to the subjects perception of cost. Subjects medical records will be reviewed for reported side affects and compared to subject reported satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Elizabeth Healthcare, Covington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes